CLINICAL TRIAL: NCT04946279
Title: Improving Decision-Making Encounters in Lung Cancer (I DECide): A Low-Literacy Conversation Tool
Brief Title: Decision Aid for the Improvement of Decision-Making in Patients With Non-small Cell Lung Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Oregon Health and Science University (Other); ATS Foundation (Unknown); Hildegard Lamfrom Endowment (Unknown); Medical Research Foundation, Oregon (Other)
Responsible Party: Principal Investigator, Donald R Sullivan, MD, MA, MCR, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00020688; NCI-2021-05887 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00020688 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2021-06-23; First posted 2021-06-30 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Lung Non-Small Cell Carcinoma; Stage I Lung Cancer AJCC v8; Stage II Lung Cancer AJCC v8; Stage III Lung Cancer AJCC v8; Stage IV Lung Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Practice Guidelines as Topic; Standard of Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (conversation tool) (Experimental): Patients receive the conversation tool.
  Interventions: Other: Informational Intervention; Other: Questionnaire Administration
- Arm II (usual care) (Active Comparator): Patients receive usual care.
  Interventions: Other: Best Practice; Other: Questionnaire Administration

INTERVENTIONS:
Other: Best Practice — Receive usual/standard of care
  Other Names: standard of care; standard therapy
  Arms: Arm II (usual care)
Other: Informational Intervention — Receive conversation tool
  Arms: Arm I (conversation tool)
Other: Questionnaire Administration — Ancillary studies - Baseline and follow-up questionnaires

SUMMARY:
This clinical trial refines and tests the effect of a decision aid in improving decision-making in patients with non-small cell lung cancer. Patients with cancer want to be informed about their diagnoses, treatment procedures and goals of treatment. They also seek active roles in decision-making. Shared decision-making (SDM) is the process of clinician and patient jointly participating in a health decision after discussing the options, benefits and harms, and considering the patient's values, preferences, and circumstances. SDM can improve patient involvement in decision making, satisfaction, health care quality, and quality of life. Decision aids can improve patient knowledge, create more realistic outcome expectations; reduce decisional conflict, distress, depression and uncertainty; and improve physician-patient communication and quality of life, compared with no decision aid. This trial's main aim is to evaluate the feasibility and efficacy of a decision aid in patients with non-small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Refine a conversation tool among patients with lung cancer by conducting prototype testing in an iterative process.

II. Conduct a trial at two comprehensive cancer treatment centers representing academic and Veterans Affairs medical centers.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive the conversation tool.

ARM II: Patients receive usual care.

Patients in both arms are followed up within 4-8 weeks after baseline to complete a second questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* PART I: Completed treatment for suspected or confirmed stage I-IV non-small cell lung cancer (NSCLC)
* PART I: English fluency
* PART II: Undergoing diagnostic work-up for suspected stage I-IV NSCLC
* PART II: English fluency
* PART II: > 6-month life expectancy
* PART II: Score of > 3 on the 6-Item Screener for Cognitive Impairment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2020-08-07 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the conversation tool | At enrollment
  The number of patients enrolled divided by the number of patients offered enrollment.
Acceptability of the conversation tool | At enrollment
  The number of participants who completed the conversation tool divided by the number of participants who began the conversation tool.

SECONDARY OUTCOMES:
Anxiety | From enrollment to the end of follow-up at 8 weeks
  Assessed using the Hospital Anxiety and Depression Scale.
Decisional conflict | At the end of follow-up at 8 weeks
  Assessed using the Decisional Conflict Scale.
Decisional Regret | At the end of follow-up at 8 weeks
  Assessed using the Decisional Regret Scale.
Perceived involvement in care | At the end of follow-up at 8 weeks
  Assessed using the Perceived Involvement in Care Scale.
Shared decision-making quality | At the end of follow-up at 8 weeks
  Assessed using the Shared Decision Making Questionnaire.
Decision making involvement | From enrollment to the end of follow-up at 8 weeks
  Assessed using the Control Preferences Scale.
Self-efficacy | From enrollment to the end of follow-up at 8 weeks
  Assessed using the Decision Self-Efficacy Scale.
Values-treatment concordance | From enrollment to the end of follow-up at 8 weeks
  Assessed using electronic medical record (EMR).

CONTACTS AND LOCATIONS:
Overall Officials: Donald Sullivan, Principal Investigator — OHSU Knight Cancer Institute
Locations (2):
- United States (2):
  - OHSU Knight Cancer Institute, Portland, Oregon
  - Portland VA Medical Center, Portland, Oregon